CLINICAL TRIAL: NCT06414980
Title: Examining the Effect of the Suggestion Given to Patients With the Olfactory Memory Method Before the Surgical Operation on the Vital Signs and Systemic Evaluation Scoring During Awakening.
Brief Title: Smell Memory Method for Patients Before Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, Mükremin Taşkın, Principal Investigator, Ataturk University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: B.30.2.ATA.0.01.00/688
Record Dates: First submitted 2024-05-10; First posted 2024-05-16 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Surgery; Gallbladder; Smell
MeSH Terms: conditions — Anosmia

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): On the day of the operation, patients will be given a menthol scent before the surgery. Data collection forms will be applied to the experimental group at specified intervals on the day of operation, at the clinic exit, before surgery, after surgery and in the recovery room (PACU). The day after the operation, a final interview will be held with the experimental group patients and questions will be asked about their experiences during the post-operative awakening process and these will be recorded.
  Interventions: Behavioral: Experimental
- Control (No Intervention): In the control group, which did not undergo any intervention, at the clinic exit on the day of the operation, vital values (pulse, blood pressure) were recorded at preoperative, postoperative and recovery room (PACU) intervals (Unit entrance, 5th minute, 10th minute, 15th minute and 20th minute). , body temperature, blood pressure and SpO2) will be taken. At the same time, the Modified Aldrete Score (MAS) and the Alertness and Sedation Observer Rating Scale (OSS/S) will be independently evaluated and recorded by the researcher.

INTERVENTIONS:
Behavioral: Experimental — The effect of suggestion given to patients with the olfactory memory method before the surgical operation on vital signs and systemic evaluation scoring during awakening.
  Arms: Experimental

SUMMARY:
The research is planned as a randomized controlled experimental at Erzurum Atatürk University Health Application and Research Center.

The population of the research will include patients who come to the General Surgery Gastroenterology service for laparoscopic cholecystectomy between the specified dates and who meet the criteria for inclusion in the study. In this research, 30 experimental and 30 control group patients will be included in the study in order to perform parametric tests.

The data of the research were prepared by the researcher using the literature and similar studies after obtaining ethics committee approval and written permission from the institution where the research would be conducted. "FR.3- Alertness and Sedation Observer Assessment Scale (OAA/S)" and Modified Aldrete Scoring, Awake and Sedation Observer Assessment Scale and "FR.4- MAS and OAA/S Scores Time-Dependent", which includes the Patient's Vital Signs, are used to evaluate the patient's condition. Patients determined by the "Change Table" will be collected by observing them before and after surgery.

In the research; In order to more easily overcome the anxiety and confusion that patients who have undergone surgical operations experience during the orientation process while waking up after the case, the patient will be given suggestions regarding the post-anesthesia waking period by testing the menthol smell in the preoperative period. When the patient hears the menthol scent applied during postoperative awakening; It is intended for the patient to remember that his surgery is over, that he needs to wake up and that the medical staff is waiting for him to wake up. In this way, it is thought that the patient's anxiety and complexity during the postoperative awakening period will be eliminated, the patient's vital signs will remain at an optimum level, and a more comfortable reanimation will occur.

ELIGIBILITY:
Inclusion Criteria:

* Students who do not have communication barriers or hearing, speaking or perception problems will participate in the research.
* Those who are over 18 years of age and under 80 years of age,
* Will participate in the study voluntarily,
* Those who will undergo elective laparoscopic cholecystectomy surgery,
* Operation duration of 1 hour or more,
* General anesthesia will be applied,
* Patients without chronic loss of smell

Exclusion Criteria:

* Those who do not accept to work,
* Having problems in smelling,
* Emergency surgeries that occur outside the daily surgery list

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-06-01 (Estimated); Study Completion 2024-07 (Estimated)

PRIMARY OUTCOMES:
Modified Aldrete Score | 1 day
  The Aldrete score was first described in 1970 by Dr Antonio Aldrete as an analogue of Apgar scoring. This scoring system examines muscle activity, respiration, blood pressure, consciousness and skin color, with each given 0, 1 or 2 points, giving a maximum score of 10. Patients with a total score of 8 or above can be easily sent from the recovery room. The Modified Aldrete Scoring has become widely accepted in assessing postanesthetic recovery. It has been widely used in many postanesthesia care units41 since its description. When the Modified Aldrete Score is calculated as 9 or above, it indicates that patients are adequately prepared for transfer from the postanesthesia care unit to the service. Today, organizations such as the Canadian Association of Anesthesiologists, the Joint Commission on Accreditation of Healthcare Organizations, and the Ontario Perianesthesia Nurses Association recommend the use of the Modified Aldrete Scoring.

SECONDARY OUTCOMES:
Observer Rating of Alertness and Sedayson Scale (OSS/S) | 1 day
  The Alertness and Sedation Observer Assessment Scale (OAA/S) is a scoring system used to evaluate the alertness state in patients. In today's anesthesia practices, the OAA/S score is widely used to evaluate the level of consciousness suppression of hypnotic drugs and the alertness of patients.
  The OAA/S score was first introduced by Chernik et al. in 1990. This scoring system is an evaluation based on scoring the patient's response between 0-5. The patient's reaction status is examined, starting with calling the patient in a normal tone of voice, progressing to light poking and shaking, and if necessary, giving painful stimuli (squeezing the trapezius). Patients with scores of 5-4-3 are considered responsive, while patients with scores of 0-1 are considered unresponsive. Patients with scores between 2 and 3 are considered to have loss of consciousness.

CONTACTS AND LOCATIONS:
Locations (1):
- Mükremin Taşın, Erzurum, Turkey (Türkiye)